CLINICAL TRIAL: NCT05282147
Title: Can the Diagnostic Accuracy of Newborn Eye Screening for Congenital Cataract be Improved With Digital Dual Light Source Imaging? The Digital Imaging vs Ophthalmoscopy (DIvO)Study.
Brief Title: Digital Imaging Versus Ophthalmoscopy
Acronym: DIvO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Louise Allen, Chief Investigator, Cambridge University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CCTU0276
Record Dates: First submitted 2022-03-08; First posted 2022-03-16 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Congenital Cataract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Babies undergoing newborn eye screening (Other): Babies having newborn eye screening with the intervention (Digital Imaging) technique in addition to the standard ophthalmoscopic technique.
  Interventions: Device: Neocam

INTERVENTIONS:
Device: Neocam — Screening within 72 hours of birth will be completed using the digital imaging device Neocam which painlessly images the eye's reflection firstly to infrared light and then to a brief green light flash.

SUMMARY:
Cataract (cloudiness of the lens) is the major cause of avoidable child blindness in the world and affects 1 in 3000 UK infants. Screening may fail to detect a cataract in an affected child (false-negative) or mistakenly suggest there is a cataract (false positive) triggering urgent unnecessary referral.

Screening is currently undertaken using an ophthalmoscope into the eye to assess the reddish reflected light (red-reflex). This study aims to test if screening using a new hand-held digital imaging device (Neocam) is more accurate than the ophthalmoscope for newborn eye screening.

DETAILED DESCRIPTION:
Cataract (cloudiness of the lens) is the major cause of avoidable child blindness in the world and affects 1 in 3000 UK infants. Cataracts are present in both eyes in more than half of the babies affected. Surgery is required by 8 weeks of age to prevent permanent visual impairment at this critical time of vision and brain development. All UK babies are examined (screened) for cataract twice within the first 8 weeks of life but late diagnosis continues to be a problem, causing avoidable visual impairment in some affected children.

Screening may fail to detect a cataract in an affected child (false-negative) or mistakenly suggest there is a cataract (false positive) triggering urgent unnecessary referral, parental anxiety and wasted NHS resources. Screening is currently performed by midwives and doctors shining a bright white light torch (an ophthalmoscope) into the eye to assess the reddish reflected light (red-reflex), similar to "red eye" seen in flash photos. Cataract causes a dark shadow on the red-reflex but the test can be difficult because bright light causes the pupils to constrict and the babies to forcefully shut their eyes. Assessment is particularly difficult in ethnic minority infants since eye pigmentation affects the hue and brightness of the red-reflex.

This study aims to test if screening using a new hand-held digital imaging device (Neocam) is more accurate than the ophthalmoscope for newborn eye screening. Neocam painlessly images the eye's reflection firstly to infrared light and then to a brief green light flash. Its infrared light causes no pupil constriction or avoidance response and the reflection is bright and consistent regardless of the baby's ethnicity. Its brief green flash and immediate imaging allows a photo of the red-reflex to be captured before the pupil has time to constrict.

To compare the accuracy of both tests, the investigators seek to enrol 140,000 newborn babies in a two year study period. All babies will have both the current ophthalmoscope screening test and additional Neocam imaging. If either test is potentially abnormal, the baby will be referred for specialist examination.

A more accurate screening test could prevent life-long disability and reduce costs to the NHS and society. This study will allow a future estimation of what these savings might be and whether changing to a digital imaging screening service might be justified. The result may have an impact on eye screening world-wide to prevent childhood blindness from cataract.

ELIGIBILITY:
Inclusion Criteria:

All newborn babies having the newborn physical examination

Exclusion Criteria:

None

Max Age: 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140000 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the screening evaluation of the Neocam (intervention) test | 2 years
  The proportion of patients correctly identified as having cataract by a positive Neocam screening test result. Where a higher value indicates better sensitivity of the screening test for presence of cataract.
Specificity of the screening evaluation of the Neocam (intervention) test | 2 years
  The proportion of patients correctly identified as not having cataract by a negative Neocam screening test result. Where a higher value indicates better specificity of the screening test for absence of cataract.
Sensitivity of the screening evaluation of the standard test | 2 years
  The proportion of patients correctly identified as having cataract by a positive standard screening test result. Where a higher value indicates better sensitivity of the screening test for presence of cataract.
Specificity of the screening evaluation of the standard test | 2 years
  The proportion of patients correctly identified as not having a cataract by a negative standard screening result. Where a higher value indicates better specificity of the screening test for absence of cataract.

SECONDARY OUTCOMES:
Usability feedback | 2 years
  Qualitative usability feedback and test preference using screener questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Allen, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust